CLINICAL TRIAL: NCT03225235
Title: Prospective Evaluation of Hypofractionated Stereotactic RT (SBRT) Using CyberKnife for Patients With Low and Intermediate Risk of Progression Prostate Cancer.
Brief Title: Prospective Evaluation of Hypofractionated Stereotactic RT Using CyberKnife for Patients With Prostate Cancer
Acronym: CYBERPROST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYBERPROST
Record Dates: First submitted 2017-05-19; First posted 2017-07-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer, SBRT, Ultrafractionation, CyberKnife
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Stereotactic SBRT (Experimental): By assuming a hypofractionated irradiation scheme, it is assumed that between the fractions sublethal radiation damage is being treated and the time factor does not significantly affect RT result. The SBRT fractional dose was determined on the basis of a Biologically Effective Dose (BED) calculation using a linear-square model, which assumes that α / β takes the following values for:
  * tumor (RS) = 1.5
  * Late rectal and bladder complications = 3.0
  * early rectal and bladder complications = 10.0.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — hypofractionated stereotactic radiotherapy (SBRT) using CyberKnife for Patients With Low and Intermediate Risk of Progression Prostate Cancer

SUMMARY:
The main purpose of study is to evaluate hypofractionated stereotactic radiotherapy (SBRT) using CyberKnife for Patients with low and intermediate risk of progression prostate cancer.

DETAILED DESCRIPTION:
Evaluation of the usefulness expression of selected proteins (PTEN, SMAD4, Cyclin D1, SPP1) as prognostic and predictive factors.

ELIGIBILITY:
Inclusion Criteria:

* men from 40 to 75 years of age with a confirmed adenocarcinoma prostate, prostate biopsy will be performed <180 days prior to the randomization date,
* completed assessment of tumor differentiation according to Gleason grading allows to perform stratification;
* general Performance Status according to the Eastern Cooperative Oncology Group (ECOG) classification ( 0 -1),
* belonging to the group of low and intermedium risk of progression; (cT1-cT2c, Gleason 7, PSA to 19.9 ng / ml), cT specified by AJCC 7 Edition (appendix 2),
* PSA marked at least 10 days after or before the biopsy, and for patients taking phytosterol 30 days after discontinuation,
* no distant metastases,
* signing informed consent,
* morphological and biochemical blood parameters within the normal limits.

Exclusion Criteria:

* the presence of active cancer, except skin cancer preceding period 5 years prior to randomization,
* surgical treatment (radical prostatectomy) or RT in the pelvic area,
* co-morbidities that may significantly affect the expectancy life of the patients
* do not meet the criteria for inclusion.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-08-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
survival time without biochemical recurrence, | 5 years
  Phoenix definition of biochemical failure

SECONDARY OUTCOMES:
survival time specific for prostate cancer, | 5 years
  the period of time from randomization until death from prostate cancer

OTHER OUTCOMES:
QoL-EORTC quality of life | 5 years
  For QoL the EORTC questionnaire (C30 with PR25) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Milecki, PhD., MD, Principal Investigator — Greater Poland Cancer Centre
Locations (1):
- Greater Poland Cancer Centre, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes